CLINICAL TRIAL: NCT00650585
Title: Promising Programs for Substance Abuse Prevention: Replication and Evaluation Initiative
Brief Title: An Effectiveness Trial of Project ALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2003-DR-FX-001; 2007-JF-FX-0064 (Other Grant/Funding Number: Dept. of Justice, OJJDP)
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Alcohol Drinking; Smoking; Marijuana Smoking
Keywords: smoking; alcohol; prevention; prevention & control
MeSH Terms: conditions — Alcohol Drinking; Smoking; Marijuana Smoking | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Did not receive Project ALERT
- Treatment group (Experimental): Received Project ALERT
  Interventions: Behavioral: Project ALERT

INTERVENTIONS:
Behavioral: Project ALERT — Project ALERT (Adolescent Learning Experiences in Resistance Training) is a drug prevention curriculum designed for middle-school students (11 to 14 years old). The 11 lessons in the first year and 3 booster lessons in the second year focus on alcohol, tobacco, marijuana, and inhalants - the substances that adolescents are most likely to use. Project ALERT uses participatory activities and videos to help motivate youth to avoid drug use, to teach youth skills and strategies to resist peer pressures to use drugs, and to establish social norms against drug-use. More information about Project ALERT may be found at http://www.projectalert.best.org/.
  Other Names: Adolescent Learning Experiences in Resistance Training
  Arms: Treatment group

SUMMARY:
The purpose of this study is to replicate a longitudinal evaluation of Project ALERT, a substance abuse prevention program that targets middle school students.

DETAILED DESCRIPTION:
Project ALERT is a substance abuse prevention program that targets middle school students. The purposes of this evaluation are to test its immediate and one-year effectiveness in a randomized experimental design that will span a total of 2.5 years for each of two cohorts. The cohorts are spaced one year apart to reduce our implementation and data collection burdens at any one time. The design for the two cohorts is identical. In schools randomly assigned to the treatment group, instructors receive Project ALERT training and materials prior to beginning the program and have access to technical assistance on request. In schools randomly assigned to the control group, teachers implement whatever substance abuse prevention curricula they normally would (if any).

ELIGIBILITY:
Inclusion Criteria:

* schools with 6th-8th grades housed together on a common campus
* schools with 6th grade student population of at least 100 students
* schools with no current 6th, 7th, or 8th grade implementation of any drug prevention curriculum recognized as a model program by a federally-sponsored registry
* all regular education students in the targeted grade must participate

Exclusion Criteria:

* students in self-contained classrooms (i.e., special education classes)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8338 (Actual)
Dates: Start 2004-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris L Ringwalt, DrPH, Principal Investigator — Pacific Institute for Research & Evaluation; Heddy K Clark, Ph.D., Study Director — Pacific Institute for Research & Evaluation
Locations (1):
- Pacific Institute for Research & Evaluation, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Ringwalt CL, Clark HK, Hanley S, Shamblen SR, Flewelling RL. Project ALERT: a cluster randomized trial. Arch Pediatr Adolesc Med. 2009 Jul;163(7):625-32. doi: 10.1001/archpediatrics.2009.88. PMID 19581545
- See also: Project ALERT website — http://www.projectalert.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Schools with grades 6-8 who did not currently use an evidence-based substance use prevention program in those grades, and committed themselves to including all their sixth grade students were recruited. Schools were recruited in two cohorts spaced one year apart (2004-2005 and 2005-2006 academic years). Schools from 11 states were enrolled.
Groups:
- Control Group: School did not receive Project ALERT, a substance use prevention program
- Treatment Group: School received Project ALERT, a substance use prevention program with 11 lessons the first year and 3 booster lessons the second year
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 4348 | 3990
Completed | 2551 (Completed posttest--a self-report survey administered 30 approximately 30 days after treatment) | 2513 (Completed posttest--a self-report survey administered 30 approximately 30 days after treatment)
Not Completed | 1797 | 1477
Not completed — Lost to Follow-up | 505 | 482
Not completed — No parental consent | 935 | 866
Not completed — Excluded/ruled ineligible | 357 | 129

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 4348 | 3990 | 8338
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4348 | 3990 | 8338
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2178 | 2051 | 4229
  Male | 2170 | 1939 | 4109

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 30-day Use of Alcohol
Description: Students completed an 81-item self-report questionnaire. They were asked on how many days they had used alcohol in the previous 30 days. Response options included "none," "1 or 2 days in the last month," "3 to 5 days in the last month," "6 to 19 days in the last month," and "20 or more days in the last month." Response options were dichotomized into none and at least one day.
Time Frame: measured approximately 30 days after intervention completed
Population: Data were cleaned to remove cases with logical inconsistencies which decreased our sample by 3.6% of respondents at pretest and 7.5% at post-test. Missing covariate data were imputed using the Expectation Maximization (EM) algorithm. Missing data were imputed using the EM algorithms implemented in the Missing Value Analysis module in SPSS 13.0.
Measure: Number; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
Participants | 330 | 332

2. Primary Outcome: Self-reported 30-day Use of Cigarettes
Description: Students completed an 81-item self-report questionnaire. They were asked on how many days they had smoked cigarettes in the previous 30 days. Response options included "none," "1 or 2 days in the last month," "3 to 5 days in the last month," "6 to 19 days in the last month," and "20 or more days in the last month." Response options were dichotomized into none and at least one day.
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 130 | 144

3. Primary Outcome: Self-reported 30-day Marijuana Use
Description: Students completed an 81-item self-report questionnaire. They were asked on how many days they had used marijuana in the previous 30 days. Response options included "none," "1 or 2 days in the last month," "3 to 5 days in the last month," "6 to 19 days in the last month," and "20 or more days in the last month." Response options were dichotomized into none and at least one day.
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 130 | 116

4. Primary Outcome: Self-reported 30-day Inhalant Use
Description: Students completed an 81-item self-report questionnaire. They were asked on how many days they had used inhalants in the previous 30 days. Response options included "none," "1 or 2 days in the last month," "3 to 5 days in the last month," "6 to 19 days in the last month," and "20 or more days in the last month." Response options were dichotomized into none and at least one day.
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 224 | 239

5. Primary Outcome: Self-reported Lifetime Alcohol Use
Description: Students completed an 81-item self-report questionnaire. To assess lifetime use, we asked if the respondent had ever used alcohol (yes or no).
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 1236 | 1288

6. Primary Outcome: Self-reported Lifetime Cigarette Use
Description: Students completed an 81-item self-report questionnaire. To assess lifetime use, we asked if the respondent had ever smoked cigarettes (yes or no).
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 439 | 544

7. Primary Outcome: Self-reported Lifetime Marijuana Use
Description: Students completed an 81-item self-report questionnaire. To assess lifetime use, we asked if the respondent had ever used marijuana (yes or no).
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 238 | 265

8. Primary Outcome: Self-reported Lifetime Inhalant Use
Description: Students completed an 81-item self-report questionnaire. To assess lifetime use, we asked if the respondent had ever used inhalants (yes or no).
Time Frame: measured approximately 30 days after intervention completed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 2358 | 2324
participants | 342 | 379

ADVERSE EVENTS:
Time Frame: 3 years
Description: This was a self-report survey. No adverse events were reported
Arm/Group | Control Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All reports and products must be submitted for review prior to publication.